CLINICAL TRIAL: NCT05540106
Title: Impact of Art Therapy on Self-Reported Pain and Anxiety Scores of Patients Waiting to Be Seen in the Emergency Department
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Lauren Marie Maloney, Clinical Assistant Professor of Emergency Medicine, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-00088
Record Dates: First submitted 2022-09-10; First posted 2022-09-14 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Anxiety; Pain
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: This is a randomized, four-armed prospective interventional study that will test the effect of nature-based coloring activities on patients' pain and anxiety scores during their ED visit. The study will consist of three intervention groups and one active control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Blank Paper and Pencil (Active Comparator)
  Interventions: Behavioral: Blank Paper and Pencil
- Nature Coloring Packet (Experimental)
  Interventions: Behavioral: Nature Coloring Packet
- Geometric Shape Coloring Packet (Experimental)
  Interventions: Behavioral: Geometric Shape Coloring Packet
- Activity Book (Experimental)
  Interventions: Behavioral: Activity Book

INTERVENTIONS:
Behavioral: Nature Coloring Packet — Coloring packet containing nature scenes
  Arms: Nature Coloring Packet
Behavioral: Geometric Shape Coloring Packet — Coloring packet containing geometric shapes
  Arms: Geometric Shape Coloring Packet
Behavioral: Activity Book — Pages containing word searches, connect the dots, etc.
  Arms: Activity Book
Behavioral: Blank Paper and Pencil — Blank sheets of paper and a pencil.
  Arms: Blank Paper and Pencil

SUMMARY:
The objective of this research is to assess the effects of engaging in coloring activities on patients' self-reported pain and anxiety scores while they wait to be seen by a physician in an emergency department (ED). The current literature on patient visits in the ED highlights the significance of anxiety, stress, and frustration in patient experiences, especially when accounting for long wait times before the physician-patient encounter. The study will address this common problem by looking at the potential impact of nature-themed or geometric shape coloring activities on the ED patient experience as it relates to self-reported anxiety and pain scores. Given that long wait times are increasingly being reported across the country, this study may offer a possible meaningful low-budget, low-resource intervention which could be offered to patients.

ELIGIBILITY:
Inclusion Criteria:

* Triage Pain Score > 3
* Age >18
* Able to provide informed consent
* English-speaking
* without concern for aggressive behavior
* Glasgow Coma Scale (GCS) of 15
* Hospital Anxiety and Depression Scale-Anxiety (HADS-A) Score > 6

Exclusion Criteria:

* Concern for aggression risk, including active concern for suicidal or homicidal ideations
* Glasgow Coma Scale (GCS) <15
* triage acuity requiring critical care evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale-Anxiety (HADS-A) Score | 8 hours
  Change in self-reported Hospital Anxiety and Depression Scale-Anxiety (HADS-A) Score following art therapy intervention (0-21, 21 = most anxious)
Numerical Pain Score | 8 hours
  Change in self-reported numerical pain score following art therapy intervention (0-10, 10 = the worst pain)

SECONDARY OUTCOMES:
Color Selection | 8 hours
  Correlation between Hospital Anxiety and Depression Scale-Anxiety (HADS-A) Score or pain score and colors selected by patient to use during art therapy
Patient impression of activities | 8 hours
  Patient engagement (reported time packet used, recommendation for others to use)

CONTACTS AND LOCATIONS:
Locations (1):
- Stony Brook University Hospital, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No